CLINICAL TRIAL: NCT06105008
Title: An Randomized, Open-label, Multicenter Phase 2 Study Comparing the Efficacy and Safety of Disitamab Vedotin With Toripalimab Verus Disitamab Vedotin Monotherapy in Subjects With Endocrine-resistant Hormone Receptor-positive, HER2-Low Unresectable Locally Advanced or Metastatic Breast Cancer
Brief Title: Study of Disitamab Vedotin With Toripalimab Verus Disitamab Vedotin in Hormone Receptor Positive, HER2-low Locally Advanced or Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the company's strategic adjustment (non-security related)
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C033
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2023-10

CONDITIONS: Breast Neoplasms
Keywords: HR+breast cancer; HER2-low breast cancer; advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — disitamab vedotin; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disitamab Vedotin + Toripalimab (Experimental): Disitamab Vedotin（RC48-ADC）with Toripalimab （JS001）arm
  Interventions: Drug: Disitamab Vedotin; Drug: Toripalimab
- Disitamab Vedotin (Active Comparator): Disitamab Vedotin（RC48-ADC） arm
  Interventions: Drug: Disitamab Vedotin

INTERVENTIONS:
Drug: Disitamab Vedotin — 2.0 mg/kg intravenous (lV) infusion every 2 weeks
  Other Names: RC48-ADC, DV
Drug: Toripalimab — 3.0 mg/kg intravenous (lV) infusion every 2 weeks
  Other Names: JS001
  Arms: Disitamab Vedotin + Toripalimab

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of RC48-ADC with JS001 compared with RC48-ADC in endocrine-resistant hormone receptor (HR) positive, human epidermal growth factor receptor (HER)2-low advanced breast cancer.

DETAILED DESCRIPTION:
Eligible patients will be those patients who have had disease progression on at least 1 previous line of endocrine therapies given for the treatment of metastatic disease or relapsed within 12 months of the end of adjuvant endocrine therapy or during adjuvant endocrine therapy, patients treated with CDK4/6 inhibitors require ≥50%. All patients must have historically confirmed HR positive, HER2-low (defined as IHC2+/ISH- and IHC 1+) expression, as determined by central laboratory testing results, advanced breast cancer. IHC 1+ account for no more than 60% The study aims to evaluate the efficacy, safety and tolerability of RC48-ADC with JS001 compared with RC48-ADC. This study aims to see if RC48-ADC with JS001 allows patients to live longer without the cancer getting worse, compared to patients receiving RC48-ADC. This study is also looking to see how the treatment and the cancer affects patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older years at the time of consent
2. Pathologically confirmed breast cancer
3. Stage III unresectable locally advanced or stage IV metastatic breast cancer.
4. Subjects must be willing and able to provide recent non-previously radiotherapy metastases lesions (if feasible and available) to the sponsor-designated central laboratory prior to treatment initiation or, if not feasible or available, tumor tissue blocks (or fresh tissue sections, see laboratory manuals) obtained from locally recurrent lesions for biomarker analysis, including HER2 expression and HR status. If archival tissue is not available, then a newly-obtained baseline biopsy of an accessible tumor lesion is required within 28 days prior to Cycle 1 Day 1. Biopsy must provide adequate tissue for analysis.
5. Subjects must have HER2 low expression (defined as IHC 1+ or IHC 2+/ISH-) and HR+ status (defined as recent tumor showing ER and/or PR expression ≥1% [according to ASCO/CAP 2020 guidelines]) determined by the central laboratory.
6. The subject must meet all of the following criteria:

   1. must not have received prior chemotherapy (including ADC) in the unresectable locally advanced or metastatic disease setting
   2. have undergone endocrine therapy, or patients with weak ER-positivity (1 to 10% nuclear positivity) were eligible if they were not candidates for endocrine therapy after an adequate assessment by the investigator

      * disease recurrence or progression during adjuvant endocrine therapy period or within 12 months after completion of adjuvant endocrine therapy, either alone or in combination with CDK4/6 inhibitors, OR
      * received prior endocrine therapy with documented disease progression during treatment period or thereafter in the unresectable locally advanced or metastatic disease setting, either alone or in combination with CDK4/6 inhibitors
7. An Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 assessed within 7 days prior to randomization.
8. Measurable disease as defined in RECIST v1.1
9. The following baseline laboratory data indicating adequate organ function:

   1. ANC ≥1,500/µL
   2. platelet count ≥100,000/μL
   3. hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L
   4. total bilirubin ≤1.5 × upper limit normal (ULN) OR direct bilirubin ≤ULN for subjects with total bilirubin >1.5 × ULN. Serum bilirubin ≤3× ULN for subjects with Gilbert's disease
   5. CrCl ≥40 mL/min (measured by the Cockcroft-Gault formula as applicable, or 24-hour urine).
   6. ALT and AST ≤2.5× ULN without liver metastases or ≤5× ULN with liver metastases
   7. International normalized ratio (INR) or prothrombin time (PT) ≤1.5× ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
10. Subjects of childbearing potential under the following conditions:

    1. Must have a negative serum pregnancy test (minimum sensitivity 25 mIU/mL or equivalent units of beta human chorionic gonadotropin [β-hCG]) result within 7 days prior to the first dose of RC48-ADC. Subjects with false positive results and documented verification that the subject is not pregnant are eligible for participation.
    2. Must agree not to try to become pregnant during the study and for at least 4 months for subjects after the final dose of study drug.
    3. Must agree not to breastfeed or donate ova, starting at time of informed consent and continuing through 4 months for subjects after the final dose of study drug.
    4. If sexually active in a way that could lead to pregnancy, must consistently use at least 2 acceptable methods of birth control (contraception), at least one of which must be highly effective through at least 4 months for subjects after the final dose of study drug.
11. Subjects who can get someone pregnant (as defined in Section 10.4) under the following conditions:

    1. Must agree not to donate sperm starting at time of informed consent and continuing through at least 4 months after the final dose of RC48-ADC.
    2. If sexually active with a person of childbearing potential in a way that could lead to pregnancy, must consistently use at least 2 acceptable methods of birth control (contraception), at least one of which must be highly effective starting at time of informed consent and continuing through at least 4 months after the final dose of RC48-ADC.
    3. If sexually active with a person who is pregnant or breastfeeding, must consistently use a condom starting at time of informed consent and continuing through at least 4 months after the final dose of RC48-ADC.
12. The subject must provide documented informed consent.

Exclusion Criteria:

1. Known hypersensitivity to any excipient contained in the drug formulation of RC48-ADC, or pembrolizumab.
2. Prior anti-HER2 therapy, including an ADC.
3. Prior MMAE-containing agent
4. Prior immunotherapy including anti-PD-(L)1 or anti-PD-(L)2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CD137, CTLA-4, OX-40) in the LA/m setting ([neo]adjuvant anti-PD-(L)1 is allowed if last dose is ≥12 months prior to recurrence or progression).
5. History of another malignancy within 3 years prior to screening, with the exception of those with a negligible risk of metastasis or death (eg, approximate 5-year OS of ≥90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
6. Subjects with known active CNS or leptomeningeal metastasis are excluded. Subjects with definitively treated brain metastasis (surgery and/or radiotherapy) are eligible if the following criteria are met:

   1. All known CNS lesions have been treated.
   2. No evidence of clinical and radiographic disease progression in the CNS for ≥4 weeks after definitive treatment.
   3. Neurological symptoms attributed to brain metastases have returned to baseline.
   4. No utilization of steroids to manage symptoms related to CNS disease or its treatment within 14 days of randomization. Anti-convulsant therapy is allowed if the dose has been stable for 14 days.
7. Subjects with prior allogenic tissue/solid organ or bone marrow transplantation.
8. Subjects with acute, chronic, or symptomatic infections, including:

   1. Active infection requiring systemic treatment ≤7 days before dose of study drug. Routine antimicrobial prophylaxis is permitted.
   2. Known positivity for hepatitis B (HBsAg positive with HBV DNA titers above the upper limit of normal), active hepatitis C infection (positive by polymerase chain reaction [PCR] or on antiviral therapy for hepatitis C within the last 6 months). Subjects who have been treated for hepatitis C infection are permitted if they have documented sustained virologic response of 12 weeks.
   3. Known history of seropositive Human Immunodeficiency Virus.
   4. Ongoing symptomatic severe acute respiratory syndrome-associated coronavirus 2 (SARS-CoV-2) infection except for subjects who have recovered clinically but continue to have a detectable presence of SARS-CoV-2.
9. Uncontrolled cardio-cerebrovascular disease including:

   1. Cardiac failure - New York Heart Association, Class III or IV heart failure.
   2. Cardiac arrhythmia - Grade 2 or higher arrhythmia.
   3. Cardiac ischemia - unstable angina within the past 6 months, myocardial infraction or cerebral infarction within the past 6 months, etc.
   4. Hypertension - uncontrolled hypertension (systolic blood pressure >180 mmHg and/or diastolic blood pressure >100 mmHg).
   5. Other cardiovascular and cerebrovascular events (eg, pulmonary thrombosis or lower limb thrombosis) within 6 months prior to study enrollment, and the disease was assessed by the investigators to be unstable.
10. Ongoing, clinically significant toxicity (Grade 2 or higher) associated with prior anticancer treatment including systemic therapy, radiotherapy, or surgery.
11. Pre-existing neuropathy of Grade ≥2.
12. Has received prior radiotherapy within 2 weeks of start of study treatment. A subject is also excluded if radiotherapy occurred more than 2 weeks prior to start of study treatment but the subject has not recovered from radiation-related toxicities, requires corticosteroids, or has had radiation pneumonitis.
13. There are other serious lung diseases that require treatment, including but not limited to active tuberculosis, interstitial lung disease, etc.
14. Active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
15. History of (non-infectious, including radiation induced) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease.
16. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment. The use of corticosteroids for physiological replacement may be approved after consultation with the sponsor.
17. Subjects who have received anticancer treatment with chemotherapy, biologics, or investigational agents that is not completed 4 weeks prior to first dose of study treatment.
18. Treatment with any prohibited concomitant therapy.
19. Subjects who are breastfeeding, pregnant, or planning to become pregnant from time of informed consent until 4 months after final dose of study drug administration.
20. Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte-colony stimulating factors, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 4 weeks prior to study Day 1.
21. Other serious underlying medical condition, psychiatric or substance abuse disorder that, in the opinion of the investigator, would impair the subject's ability to receive or tolerate the planned treatment, or comply with the requirements of the study and follow-up.
22. Has received any live or live attenuated vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS), evaluated by investigator | Until progression or death, assessed up to approximately 36 months
  Defined as time from date of randomization until the date of objective radiological disease progression by investigator assessment according to RECIST v1.1 or death.

SECONDARY OUTCOMES:
Overall survival (OS) | Until death, assessed up to approximately 36 months
  Defined as the time from randomization to death due to any cause
Objective Response Rate (ORR) | Until progression, assessed up to approximately 36 months
  Defined as the percentage of patients with at least one visit response of complete or partial response (CR or PR) by Investigator assessment according to RECIST v1.1.
Disease Control Rate (DCR) | Until progression, assessed up to approximately 36 months
  Percentage of patients with complete response, partial response, or stable disease for a certain period of time according to RECIST v1.1.
Duration of response (DoR) | Until progression, assessed up to approximately 36 months
  Defined as the time from the date of first documented response (CR/PR) until the first progression or death in the absence of disease progression by Investigators assessment according to RECIST 1.1
Type, incidence, relatedness, severity, and seriousness of AEs | Up to follow-up period, approximately 36 months
  According to NCI-CTCAE Version 5.0 per each treatment arm
Incidence of laboratory tests abnormalities | Up to follow-up period, approximately 36 months
  To be summarized using descriptive statistics
Incidence of ECG abnormalities | Up to follow-up period, approximately 36 months
  To be summarized using descriptive statistics
Incidence of echocardiograms abnormalities | Up to two years after the last dose, approximately 36 months
  Change from baseline of LVEF
Health-related quality of life - EORTC-QLQ-C30 | Assessed up to approximately 36 months
  Change from baseline in the physical functioning subscale of the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) scores. Scale scores range from 0-100. For functioning and global health status/ QoL scales, higher scores indicate better functioning or global health status/QoL. For symptom scales, higher scores indicate greater symptom burden

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Fang, Ph.D, Study Director — RemeGen Co., Ltd.
Locations (3):
- China (3):
  - Binghe Xu, Beijing, Cancer Hospital Chinese Academy of Medical Sciences
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Hunan Cancer Hospital, Changsha

IPD SHARING:
Plan to Share IPD: No